CLINICAL TRIAL: NCT06964451
Title: Assessing the Effect of Virtual Reality Gamification on Anxiety and Pain Management During Extraction of MIH-affected Lower First Permanent Molars in Pediatric Patients
Acronym: VRGAMIFICATION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rasa Mladenovic (Other)
Responsible Party: Sponsor-Investigator, Rasa Mladenovic, Assistant professor, Pediatric dentist, University of Kragujevac
Organization: University of Kragujevac (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 01-14788/2022; Ethics Committee (Other: Faculty of Medical Sciences University of Kragujevac, Serbia)
Record Dates: First submitted 2025-04-23; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Virtual Reality; Distraction; Gamification; Tooth Extraction
Keywords: virtual reality; distraction; gamification; tooth extraction; MIH
MeSH Terms: interventions — Tooth Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NON VR (Active Comparator): In the extraction of one tooth, the procedure was performed according to the standard protocol (Non VR Phase).
  Interventions: Procedure: Extraction tooth
- VR (Active Comparator): For the tooth on the opposite side, the entire extraction procedure (including the application of local anesthesia) was conducted using a gamification model with VR goggles (VR Gamification Phase)
  Interventions: Procedure: Extraction tooth

INTERVENTIONS:
Procedure: Extraction tooth — Extraction of MIH Grade 4 molar

SUMMARY:
The aim of this study was to evaluate the effectiveness of gamified virtual reality in reducing anxiety and pain during the extraction of lower first molars with MIH under local anaesthesia.

DETAILED DESCRIPTION:
Dental anxiety can be tiggered by previous negative experiences, fear of pain, or loss of control, leading to avoidance of dental treatments and worsening oral health. To alleviate anxiety, various pharmacological and non-pharmacological measures are applied, including distraction as a cognitive-behavioral approach. One innovative method of distraction is gamification, which involves the use of Virtual Reality (VR) to redirect patients' focus to something relaxing instead of the treatment itself. The aim of this research was to evaluate the effectiveness of gamified virtual reality in reducing anxiety and pain during the extraction of molar-incisal hypomineralization (MIH) affected lower first molars under local anaesthesia. In prospective study, gamified virtual reality was applied during the extraction of lower first molars in 56 subjects using the split-mouth method. Through VR goggles, patients were immersed in a virtual video game world to distract them from the dental procedure.

ELIGIBILITY:
Inclusion Criteria:

* Indication for the extraction of both lower first molars due MIH grade 4.

Exclusion Criteria:

* Exclusion criteria for the study encompassed individuals with systemic disease, special needs, patients with a history of epileptic seizures or episodes of dizziness, as well as patients suffering from claustrophobia.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Face Scale | 1 day
  We used the Wong-Baker Face Scale to assess pain, which allows patients to visually describe their level of pain. This scale consists of six faces with different expressions, ranging from a face showing no pain to a face representing the worst possible pain. This method of assessment is particularly useful for children. Pain was recorded during the administration of anaesthesia and during the tooth extraction procedure
Heart rate | 1 day
  Additionally, heart rate was monitored to assess the patient's physiological response to stress and pain during the procedure. Heart rate was recorded during anaesthesia administration and during the procedure using a smartwatch that allows continuous heart rate tracking (Samsung Galaxy Watch). This type of measurement provides additional information on how the patient responds to pain and stress, enabling the dentist to adjust their approach according to the patient's physiological response.

SECONDARY OUTCOMES:
Satisfaction questionnaire | 1 day
  After the extraction procedure with VR application, patients filled out a modified satisfaction questionnaire. Responses were classified based on a 5-point Likert scale: 1 = strongly disagree, 2 = disagree, 3 = neutral, 4 = agree, and 5 = strongly agree. The post-clinical questionnaire included questions related to reduction of fear of anaesthesia and extraction, effectiveness of VR in diverting attention from the procedure, experience of discomfort during the procedure, enjoyment of the VR experience, and the potential of VR in overcoming fear of other procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty od Medical Sciences University of Kragujevac, Kragujevac, Serbia

IPD SHARING:
Plan to Share IPD: No